CLINICAL TRIAL: NCT06380192
Title: Developmental and Epileptic Encephalopathy of Genetic Etiology: Natural History Through Reuse of Clinical Data / DEE-RETRO
Brief Title: Developmental and Epileptic Encephalopathy of Genetic Etiology: Natural History Through Reuse of Clinical Data
Acronym: DEE-RETRO
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ22-DEE-RETRO
Record Dates: First submitted 2024-03-28; First posted 2024-04-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Developmental and Epileptic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patient inclusion criteria:
  * Diagnosis of developmental and epileptic encephalopathies
  * Affiliation with, or beneficiary of, a social security scheme
  Criteria for non-inclusion of patients:
  * Opposition of the patient or his/her parents in the case of minors to the re-use of data for this study.
  * Persons subject to a safeguard of justice measure
- Control patient: Inclusion criteria for controls:
  * Patients who, as part of their routine health care, require an EEG examination
  * Patients with sufficient follow-up to rule out a diagnosis of epilepsy, including developmental and epileptic encephalopathies
  * Enrolled in or receiving social security benefits
  Criteria for non-inclusion of controls :
  * Patient with a neurological or extra-neurological disease that may have an impact on the child's neurological development and outcome
  * Opposition of the patient or his/her parents to the re-use of data for this study
  * Persons subject to a safeguard of justice measure

SUMMARY:
Developmental and Epileptic Encephalopathy (DEE) are a heterogeneous group of neurodevelopmental disorders linked to both epilepsy and its underlying etiology, independently of epileptiform activity.

The creation of a database with retrospective follow-up of a large number of patients on a national scale will enable better knowledge of specific biomarkers, and thus a better classification and understanding of the natural evolution of DEE according to their etiology. This will enable better, more personalized therapeutic management of patients, depending on etiology and the presence or absence of these biomarkers. The investigators will also be able to draw up management recommendations, which are currently non-existent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Developmental and Epileptic Encephalopathy
* Registered with or benefiting from a social security scheme.

Exclusion Criteria:

* Opposition of the patient or his/her parents to the re-use of data in the context of this study
* Person subject to a safeguard of justice measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient diagnosed with developmental encephalopathy and epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of diagnostic and early predictive biomarkers of a neurodevelopmental trajectory with epileptic and developmental encephalopathies | Data 2002-2026
  This composite outcome includes multiple diagnostic domains (Clinical, biological, radiological, genetic and electroencephalographic variables)

SECONDARY OUTCOMES:
Identification of patient subgroups presenting the identified biomarkers | Data 2002-2026
  To identify patient subgroups, correlation analyses will be carried out to highlight any common clinical, biological, genetic, radiological and electroencephalographic findings.
Assessment of patients' quality of life | Data 2002-2026
  The SF-12 questionnaire is used to assess quality of life.
Assessment of age-related adaptive behavior | Data 2002-2026
  To assess the age of adaptive behavior, the Vineland II scale is the reference test.
Assessment of behavioral disorders | Data 2002-2026
  The CBCL (Child Behaviour Checklist) questionnaire is the reference test for assessing behavioural problems.
Assessment of autism spectrum disorders | Data 2002-2026
  The Social Communication Questionnaire (SCQ) will be used to assess autism spectrum disorders.

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - CHU Amiens, Amiens
  - CH Angers, Angers
  - Chu Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon HCL, Lyon
  - Assistance Publique Hopitaux de Marseille, Marseille
  - CHU de Nancy, Nancy
  - Hopitaux Pediatriques de Nice CHU Lenval, Nice
  - Necker-Enfants Malades Hospital, Paris
  - CHU Pitié Salpétrière, Paris
  - CHU Robert Debré, Paris
  - Hôpital Armand Trousseau, Paris
  - Chu Reims, Reims
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours
  - Hôpital André Mignot (CH Versailles), Versailles